CLINICAL TRIAL: NCT04307251
Title: Comparative Outcomes Between Imageless Robotic-assisted and Conventional Total Knee Arthroplasty : A Prospective, Randomized Controlled Trial
Brief Title: Comparative Outcomes Between Imageless Robotic-assisted and Conventional Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COA 012/2563
Record Dates: First submitted 2020-02-28; First posted 2020-03-13 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Navio™ Robotics-assisted Surgical System (Experimental)
  Interventions: Device: Navio™ Robotics-assisted Surgical System, LEGION Total Knee System
- Conventional, non-robotics-assisted total knee surgical system (Experimental)
  Interventions: Device: Conventional, LEGION Total Knee System

INTERVENTIONS:
Device: Navio™ Robotics-assisted Surgical System, LEGION Total Knee System — Robotic TKA uses computer software to convert anatomical information into a virtual patient-specific 3D reconstruction of the knee joint.The surgeon uses this virtual model to plan optimal bone resection, implant positioning, bone coverage, and limb alignment based on the patient's unique anatomy.
  Arms: Navio™ Robotics-assisted Surgical System
Device: Conventional, LEGION Total Knee System — Total Knee Arthroplasty (TKA) is a widespread orthopaedic procedure for restoring functionality and minimizing pain due to end stage osteoarthritis. Conventional TKA, well-accepted as the standard of care, is performed with manual instrumentation guided by intramedullary or extramedullary alignment rods, as well as rotational guides that are not patient-specific.
  Arms: Conventional, non-robotics-assisted total knee surgical system

SUMMARY:
The purpose of this study is to compare post-operative mechanical alignment (Hip-Knee-Ankle angle; HKA) between imageless robotic-assisted (Navio™ Robotics-assisted Surgical System) and Conventional Total Knee Arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee who were scheduled for a primary total knee arthroplasty
* Age 50-80 year
* Patients with osteoarthritis who voluntarily participated in the project

Exclusion Criteria:

* Patients with osteoporosis
* History of inflammatory arthroplathy
* Previous fracture or open surgery on the same knee
* Patients with bilateral total knee arthroplasty
* Patients osteoarthritis with revision surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Mechanical axis | Change from baseline mechanical axis at 6 weeks after surgery
  Post-operative Mechanical Alignment; Hip-Knee-Ankle angle; If you divide the knee into quadrants, the ideal mechanical axis would bisect the knee (0), with medial zone (-1) or lateral zone (-1) being within physiologic range. With the notable exception of physiologic varus <age 2 and physiologic valgus <age 6, medial or lateral zones 2 or 3 would likely manifest symptoms and gait disturbance and thereby warrant surgical intervention

SECONDARY OUTCOMES:
Knee Society and Knee Society function score | Change from baseline Knee Society and Knee Society function score at 3 months, 6 months, and 12 months after surgery
  Knee Society and Knee Society function score (minimum 0, maximum 200)
Range of motion of knee | Change from baseline Range of motion of knee at 3 months, 6 months, and 12 months after surgery
  Range of motion of knee (minimum 0, maximum 140)
Oxford knee score | Change from baseline Oxford knee score 3 months, 6 months, and 12 months after surgery
  Oxford knee score (minimum 0, maximum 48)

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand